CLINICAL TRIAL: NCT00302211
Title: A Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of the Addition of Inhaled Iloprost in Patients With Pulmonary Arterial Hypertension Receiving Oral Sildenafil
Brief Title: The "VISION" Trial: Ventavis Inhalation With Sildenafil to Improve and Optimize Pulmonary Arterial Hypertension
Acronym: VISION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to slow enrollment
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: C200-006
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Results first posted 2010-08-13 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Hypertension
Keywords: PAH; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate; Bosentan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- DB inhaled iloprost 6x/day (Experimental): inhaled iloprost (5 μg) 6 times per day (6×/day) plus sildenafil with or without bosentan during the double blind period
  Interventions: Drug: Inhaled Iloprost (5 μg); Drug: Sildenafil; Drug: Bosentan
- DB inhaled iloprost 4x/day (Experimental): Inhaled iloprost (5 μg) 4×/day plus inhaled placebo 2x/day plus sildenafil with or without bosentan during the double blind period
  Interventions: Drug: Inhaled Iloprost (5 μg); Drug: Inhaled Placebo; Drug: Sildenafil; Drug: Bosentan
- DB inhaled placebo 6x/day (Placebo Comparator): Inhaled placebo 6×/day plus sildenafil with or without bosentan during the double blind period
  Interventions: Drug: Inhaled Placebo; Drug: Sildenafil; Drug: Bosentan
- OL inhaled iloprost 6x/day (Experimental): Inhaled iloprost (5 μg) 6 times per day (6×/day) plus sildenafil with or without bosentan during the Open-Label treatment period
  Interventions: Drug: Inhaled Iloprost (5 μg)
- OL inhaled iloprost 4x/day (Experimental): Inhaled iloprost (5 μg) 4 times per day (4×/day) plus sildenafil with or without bosentan during the Open-Label treatment period
  Interventions: Drug: Inhaled Iloprost (5 μg)

INTERVENTIONS:
Drug: Inhaled Iloprost (5 μg) — iloprost inhalation solution (Ventavis) (5 μg)
  Arms: DB inhaled iloprost 4x/day; DB inhaled iloprost 6x/day; OL inhaled iloprost 4x/day; OL inhaled iloprost 6x/day
Drug: Inhaled Placebo — inhaled placebo
  Arms: DB inhaled iloprost 4x/day; DB inhaled placebo 6x/day
Drug: Sildenafil — oral sildenafil (dosage between 60 and 300 mg/day)
  Arms: DB inhaled iloprost 4x/day; DB inhaled iloprost 6x/day; DB inhaled placebo 6x/day
Drug: Bosentan — oral bosentan (dosage between 62.5 and 125 mg BID)
  Arms: DB inhaled iloprost 4x/day; DB inhaled iloprost 6x/day; DB inhaled placebo 6x/day

SUMMARY:
The purpose of this multi-center international trial is to evaluate the safety and effectiveness of adding iloprost or placebo (an inactive substance that contains no active study drug) to sildenafil therapy for pulmonary arterial hypertension (PAH). The study will also examine whether patients on sildenafil can reduce the number of iloprost inhalations from the approved 6 doses per day to 4 doses per day.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-85 years; of either gender.
* Confirmed PAH due to idiopathic pulmonary arterial hypertension (IPAH) or familial pulmonary arterial hypertension (FPAH).
* 6-minute walk distance (6-MWD) between 100-450 meters at screening.
* On a stable dose of sildenafil, with or without bosentan.

Exclusion Criteria:

* Any treatment for PAH with prostacyclins, prostacyclin analogues, endothelin-1 antagonists, or phosphodiesterase-5 (PDE-5) inhibitors other than sildenafil within the past 12 weeks.
* Pulmonary hypertension due to conditions other than those stated in inclusion criteria.
* Additional PAH medications added within the past 12 weeks.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-02-01 (Actual); Primary Completion 2007-12-01 (Actual); Study Completion 2008-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nazzareno Galie, MD, Principal Investigator — Istituto Malattie Apparato Cardio Univ di Bologna

REFERENCES:
- See also: CoTherix Clinical Development — http://www1.actelion.com/en/healthcare-professionals/products/ventavis/index.page

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to slow participant enrollment, the study was prematurely terminated, and recruitment was stopped after 67 subjects had been recruited instead of 180 initially planned (37% of the originally-planned sample size)
Groups:
- DB Iloprost 6×/Day: Inhaled iloprost (5 μg) 6×/day plus sildenafil with or without bosentan
- DB Iloprost 4×/Day: Inhaled iloprost (5 μg) 4×/day plus inhaled placebo 2x/day plus sildenafil with or without bosentan
- DB Placebo 6×/Day: Inhaled placebo 6×/day plus sildenafil with or without bosentan
- OL Iloprost 6x/Day: The subjects received inhaled iloprost(5 μg) 6 times per day plus sildenafil with or without bosentan during the 32-week open-label period
- OL Inhaled Iloprost 4x/Day: Subjects in this group received inhaled iloprost (5μg) 4x/day plus sildenafil with or without bosentan during the open-label period
Period: Double Blind Period (New Patients)
Arm/Group | DB Iloprost 6×/Day | DB Iloprost 4×/Day | DB Placebo 6×/Day | OL Iloprost 6x/Day | OL Inhaled Iloprost 4x/Day
Started | 26 (These subjects had the option to continue with the same dose of iloprost during the OL period) | 27 (These subjects had the option to continue with the same dose of iloprost during the OL period) | 14 (These subjects could receive either iloprost 4x/day or 6x/day in the OL period) | 0 | 0
Completed | 23 | 25 | 10 | 0 | 0
Not Completed | 3 | 2 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 0 | 0
Not completed — Investigator's judgement | 1 | 0 | 0 | 0 | 0
Not completed — Disease progression | 0 | 1 | 1 | 0 | 0
Period: Open Label-Patients From Double-Blind
Arm/Group | DB Iloprost 6×/Day | DB Iloprost 4×/Day | DB Placebo 6×/Day | OL Iloprost 6x/Day | OL Inhaled Iloprost 4x/Day
Started | 0 | 0 | 0 | 26 (21 patients (pts) in 6x/day DB phase & 5 patients in placebo 6x/day DB phase enrolled in OL 6x/day) | 32 (26 pts in 4x/day + placebo 2x/day DB phase & 6 pts in placebo 6x/day DB phase enrolled in OL 4x/day)
Completed | 0 | 0 | 0 | 18 | 24
Not Completed | 0 | 0 | 0 | 8 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Investigator's judgement | 0 | 0 | 0 | 1 | 0
Not completed — Disease progression | 0 | 0 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — PH requiring lung transplant | 0 | 0 | 0 | 0 | 1
Not completed — Termination of the study by the sponsor | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DB Iloprost 6×/Day | DB Iloprost 4×/Day | DB Placebo 6×/Day | Total
Number analyzed (Participants) | 26 | 27 | 14 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 17 | 9 | 49
  >=65 years | 3 | 10 | 5 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (11.95) | 56.6 (16.27) | 56.9 (11.90) | 54.8 (13.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 13 | 52
  Male | 6 | 8 | 1 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 15 | 9 | 38
  United Kingdom | 4 | 2 | 1 | 7
  Spain | 0 | 1 | 1 | 2
  Italy | 0 | 1 | 0 | 1
  Germany | 7 | 6 | 3 | 16
  Austria | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline to Week 16 in 6-Minute Walk Distance (6MWD) During the Double-blind Treatment Period
Description: The 6MWD test is a non-encouraged test, performed in a 30-meter long flat corridor, where the patient is instructed to walk as far as possible, back and forth around two cones during 6 minutes. They can slow down, rest, or stop if needed. This test is used to assess exercise capacity. The test was performed about 30 minutes after study drug administration. Any increase in the walk distance was considered improvement from baseline.
Time Frame: Day 1 and Week 16
Population: Only Participants in the double-blind treatment period were included if they received at least one dose of study drug and had at least one post-baseline efficacy measure at Week 16. Due to early study termination (about 30% of the enrollment goal) the study was severely under-powered and no accurate statistical analyses could be performed.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | DB Iloprost 6×/Day | DB Iloprost 4×/Day | DB Placebo 6×/Day
Number analyzed (Participants) | 26 | 27 | 13
Meters | 10.1 (62.15) | 29.6 (55.17) | -22.0 (124.7)

2. Secondary Outcome: Number of Subjects With WHO Functional Class (WHO FC) Improvement at Week 16
Description: This test is used to assess disease severity. Four fucntional classes (FC) are defined from FC I (no limitation of physical activity) to FC IV (inability to carry out any physical activity without symptoms). Improvement is considered when a participant changes from a higher class to a lower class.
Time Frame: Day 1 and Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DB Iloprost 6×/Day | DB Iloprost 4×/Day | DB Placebo 6×/Day
Number analyzed (Participants) | 26 | 27 | 13
Participants | 4 | 6 | 0

3. Secondary Outcome: Time to Clinical Worsening
Description: Clinical worsening is defined as one of the following: death due to worsening PAH, receipt of lung or heart-lung transplantation, or atrial septostomy, hospitalization for worsening PAH, any early discontinuation from study during the blinded or open-label phase due to worsening PAH, initiation of additional PAH-specific treatment. Due to insufficient data, time could not be assessed accurately and only number of patients with clinical worsening could be reported.
Time Frame: Week 16 and Week 48
Population: Only participants who received at least one dose of study drug and with available data at Week 16 (for the double-blind period) and at Week 48 (for the open-label period) were included in the analysis
Measure: Count of Participants; unit: Participants
Groups:
- OL Iloprost 4x/Day: The subjects received inhaled iloprost (5μg) 4 times per day plus sildenafil with or without bosentan during the 32-week open-label period
Arm/Group | DB Iloprost 6×/Day | DB Iloprost 4×/Day | DB Placebo 6×/Day | OL Iloprost 6x/Day | OL Iloprost 4x/Day
Number analyzed (Participants) | 26 | 27 | 14 | 22 | 28
Participants | 0 | 1 | 1 | 2 | 3

4. Other Pre Specified Outcome: Number of Participants With Any Adverse Events
Description: This is the overall number of participants in each group who reported at least one adverse event (i.e., any untoward medical occurrence or unfavorable and unintended sign whether or not considered related to the study drug) with an onset from the first administration of study drug up to the last study visit.
Time Frame: From Day 1 to Week 16 and Week 48
Population: Safety population: All randomiized subjects who received at least one dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | DB Iloprost 6×/Day | DB Iloprost 4×/Day | DB Placebo 6×/Day | OL Iloprost 6x/Day | OL Iloprost 4x/Day
Number analyzed (Participants) | 26 | 27 | 14 | 26 | 32
Participants | 24 | 22 | 14 | 23 | 30

5. Post Hoc Outcome: Number of Participants With Change From Baseline to Week 16 in 6-Minute Walk Test (MWT) During the Double-blind Period
Description: The number of participants in the double-blind treatment period who showed improvement or worsening in the 6-MWT - from baseline distance between 100-450 meters - was assessed for each treatment group. The 6-minute walks were measured in meters. Any increase in walk distance at Week 16 was considered improvement from baseline, any decrease was considered as deterioration from baseline.
Time Frame: Week 16
Population: Only Participants in the double-blind treatment period were included if they received at least one dose of study drug and had a post-baseline efficacy measure at Week 16.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Iloprost 6×/Day | DB Iloprost 4×/Day | DB Placebo 6×/Day
Number analyzed (Participants) | 26 | 27 | 13
Participants
  6-MWT improvement | 13 | 18 | 9
  6-MWT deterioration | 12 | 8 | 4
  No change | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: from Day 1 (Baseline) up to Week 48 (or up to 30 days after the last dose of study drug for serious adverse events)
Description: Safety was assessed on the basis of adverse events, laboratory tests, physical examination and vital signs during both the double-blind and open-label phases of the study.
Arm/Group | DB Iloprost 6×/Day | DB Iloprost 4×/Day | DB Placebo 6×/Day | OL Iloprost 6x/Day | OL Iloprost 4x/Day
Serious Adverse Events (participants affected / at risk) | 3/26 | 5/27 | 3/14 | 4/26 | 13/32
Other Adverse Events (participants affected / at risk) | 24/26 | 22/27 | 14/14 | 23/26 | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Iloprost 6×/Day (N=26) | DB Iloprost 4×/Day (N=27) | DB Placebo 6×/Day (N=14) | OL Iloprost 6x/Day (N=26) | OL Iloprost 4x/Day (N=32)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 3
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Lupus vasculitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Iloprost 6×/Day (N=26) | DB Iloprost 4×/Day (N=27) | DB Placebo 6×/Day (N=14) | OL Iloprost 6x/Day (N=26) | OL Iloprost 4x/Day (N=32)
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 0 | 0 | 2 | 0
Right ventricular failure (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 0 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 4 | 1 | 1 | 2 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 1 | 1
Oedema (General disorders) | 1 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 3 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lymph gland infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 2 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 3 | 5 | 1
Headache (Nervous system disorders) | 10 | 7 | 2 | 10 | 6
Hypogeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 2 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 3 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Dyssomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Dysuria (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 2 | 4 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 4 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 1 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Medical device implantation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Cardiovascular insufficiency (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 6 | 3 | 1 | 6 | 4
Hypotension (Vascular disorders) | 3 | 4 | 1 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Swelling (General disorders) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Primary purpose was to evaluate the efficacy of iloprost in PAH patients. Due to slow recruitment only 67 of the 180 participants planned were enrolled. Consequently efficacy results are not meaningful and no statistical analyses could be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Written permission to publish results must be obtained in advance from Actelion (formerly CoTherix). Manuscript of any proposed publication must be sent to Actelion at least 30 days in advance of the submission date. Actelion will inform in writing of any objection of specific content in the proposed publication.In addition, the institution shall either delete disclosure of all potentially patentable inventions or delay submission of the proposed publication for up to 90 days.